# Faculty of Dentistry The University of Hong Kong

Prince Philip Dental Hospital 34 Hospital Road Hong Kong



香港大學牙醫學院 菲臘牙科醫院 醫院道 34 號 香港

### INFORMATION SHEET

2<sup>nd</sup> May, 2018

#### Dear Parent,

## The effectiveness of an oral health education programme in promoting healthy oral behaviors among adolescents in Hong Kong

Researcher: Clinical Associate Professor Wong Hai Ming, Dr. Cao Wang Nan, Xiang Bilu, Professor McGrath

Adolescence is an important stage for growth and development when changes in physical and oral health status are expected. Since the School Dental Care Service delivered by Department of Health only targets children in primary schools, most adolescents ignore the importance of regular dental visits when they are promoted to secondary schools. Poor oral health status not only affects the appearance, but also leads to serious oral diseases, such as gingivitis or dental caires.

Your child is invited to take part in an oral education programme conducted by the Faculty of Dentistry, The University of Hong Kong. This programme will be conducted in your child's school during the period from August 2018 to December 2020. Before making the decision, please take time to read the following information about the purpose and content of this programme. Should you have any questions, please contact us. It is our pleasure to answer your questions.

### **Project Objectives:**

Through participating in an oral education programme, adolescents will be encouraged to develop good oral hygiene habits. The effectiveness of the oral health education programme will be evaluated through dental examinations and questionnaire.

### **Project Details:**

- 1. An oral education programme will be conducted in secondary schools;
- 2. Free dental examinations will be provided to participants twice (It will be conducted by dentists and it will take no longer than 10 minutes);
- 3. All participants will be required to fill in a questionnaire about their oral health behaviors (It will take less than 15 minutes to complete the questionnaire and it will be conducted for three times).

All the oral examinations will not bring any discomforts, risks or harms to your child. <u>Your child will receive his/her examination report and a tooth cleaning kit upon completion of all the evaluations.</u> We are also glad to offer some professional prevention or treatment recommendations. <u>In addition, your child will be granted a certificate of participation delivered by the Faculty of Dentistry, The University of Hong Kong to show our encouragement and gratitude.</u>

It is up to you to decide whether or not to participate in this programme. Your participation is totally voluntary. If you decide to participate, please sign and return the consent form, and keep this information sheet as a record. Please note that you can change your decision and withdraw at any time without giving any reasons. Any refusal or withdraw will definitely NOT affect your child's medical/dental cares that received and/or will receive in the future.

Please note that any clinical treatments will not be provided in this programme. The collected information about you/your child will be kept strictly confidential and will not be identified from our publications.

This programme has been approved by the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster. This programme will be conducted by the Faculty of Dentistry, The University of Hong Kong. If you have any questions or comments about the programme, please contact Ms. Cindy Yeung at 2859 0357 during office hours.

We are grateful for your participation. Thank you very much.

### PARTICIPANT CONSENT FORM

Re: The effectiveness of an oral health education programme in promoting healthy oral behaviors among adolescents in Hong Kong

(Researcher: Clinical Associate Professor Wong Hai Ming, Dr. Cao Wang Nan, Xiang Bilu, Professor McGrath)

- 1. I confirm that I have read and understood the information sheet for the programme and have the opportunity to ask questions.
- 2. I understand that my child's participation is totally voluntary and my child is free to withdraw at any time, without giving any reason.
- 3. I understand that any medical records of my child may be reviewed by responsible personnel of Institutional Review Board of the University of Hong Kong / Hospital Authority Hong Kong West Cluster (IRB). IRB is one of the authorized parties which have access to the subjects' records related to the study for review purpose. I give my permission for them to have access to my child's records.
- 4. I agree to take part in the programme "The effectiveness of an oral health education programme in promoting healthy oral behaviors among adolescents in Hong Kong".5. I agree to let my child, \_\_\_\_\_\_, to take part in the above programme.

| Name of Child | <br>Signature | Date |
|---------------------------------|---------------|----------|
| Name of Parents/ Legal Guardian | Signature | Date |
| Name of Researcher | <br>Signature | <br>Date |

Copies to:

Researcher's File